CLINICAL TRIAL: NCT04861987
Title: A Phase 1b Dose-escalation Study of the Safety and Pharmacokinetics of Fixed-dose PCS6422 with Escalating Doses of Capecitabine Administered Orally to Patients with Advanced, Refractory Gastrointestinal Tract Tumors
Brief Title: A Study of the Safety and PK of PCS6422 (Eniluracil) with Capecitabine in Patients with Advanced, Refractory GI Tract Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Processa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCS6422-GI-01
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Advanced Cancer; Refractory Cancer; Tumor Gastric
Keywords: Capecitabine; Eniluracil
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PCS6422 + Capecitabine (Experimental): Fixed dose of PCS6422 combined with various doses of Capecitabine administered in 14 day cycles
  Interventions: Drug: PCS6422 and capecitabine

INTERVENTIONS:
Drug: PCS6422 and capecitabine — PCS6422 is an experimental drug that, when combined with capecitabine, may make the immune response more active against cancer. Capecitabine is a commonly used oral fluoropyrimidine.

SUMMARY:
This study is an open label, multicenter study in patients who have advanced, relapsed refractory GI cancer or are not relapsed/refractory but are intolerant to other therapies who, in the judgment of investigators, are candidates for fluoropyrimidine monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Has advanced, metastatic or unresectable GI tract tumors that are refractory or intolerant to existing available therapies and for whom the investigator recommends fluoropyrimidine monotherapy.
2. Has measurable disease in accordance with Respond Evaluation Criteria in Solid Tumors (RECIST) guidelines (Version 1.1).
3. Is aged ≥18 years
4. Has not received treatment with intravenous (IV) 5 FU or oral 5 FU analogs in the 4 weeks preceding enrollment
5. Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 at study entry
6. Has adequate bone marrow, liver, and renal function as assessed by the following laboratory requirements conducted within 7 days before starting study treatment:

   1. peripheral ANC of ≥1.5 × 109/L
   2. platelet count of ≥75 × 109/L without growth factor/transfusion
   3. hemoglobin ≥8.5 g/dL without growth factor/transfusion
   4. estimated glomerular filtration rate >50 mL/min
   5. total bilirubin <2 × upper limit of normal (ULN); <5 × ULN if patient has liver metastases, biliary tract cancer; or ≤3 × ULN if the patient has Gilbert's disease
   6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <2.5 × ULN, with liver metastasis <5 × ULN
   7. international normalized ratio (INR) <1.5
7. Has a life expectancy of at least 12 weeks
8. Female patients of childbearing potential and male patients with partners capable of reproduction must agree to use an effective contraceptive method from the time of Screening through 60 days after the last dose of capecitabine
9. Females of childbearing potential must have a negative serum β human chorionic gonadotropin pregnancy test result
10. Willingly provides written, informed consent.
11. Has resolution or stabilization of acute toxicity from prior therapy to Grade <2 - except Grade 2 neuropathy
12. If patient has human immune deficiency virus (HIV) infection, it is controlled with undetectable viral load with antiretroviral treatment.
13. If patient has hepatitis C infection and received antiviral treatment, has a negative viral load at Screening
14. If patient has chronic hepatitis B infection and is receiving antiviral treatment, has a negative viral load at Screening.
15. Is willing and able to comply with all protocol required visits and assessments

Exclusion Criteria:

1. Is unable to take oral medication or malabsorption syndromes potentially interfering with medication absorption (e.g., short bowel syndrome or chronic, partial bowel obstruction)
2. Has history or presence of clinically significant abnormal 12 lead ECG results, in the investigator's opinion
3. Has current brain metastasis
4. Has prolonged QTc (with Fridericia's correction) of >480 msec in men and women performed at Screening
5. Has a history of prolonged QTc interval, ventricular tachycardia/fibrillation or significant ventricular arrhythmia, or Torsades de Pointes, or a history of ventricular ablation for arrhythmia
6. Has congenital long QT syndrome or a family history of long QT syndrome
7. Has other clinically significant cardiac disease including, but not limited to, uncontrolled angina, myocardial ischemia or infarction within 6 months, congestive heart failure >Class II per the New York Heart Association, or history of myocarditis
8. Has an electrolyte disturbance, such as uncorrected hypokalemia/hyperkalemia, hypomagnesemia, or hypocalcemia. Patients can be enrolled following successful correction of an electrolyte disturbance.
9. Is currently using any drugs included in the prohibited medications list in the protocol (including those that can prolong QTc) that cannot be discontinued
10. Has known hypersensitivity to any of the components of study treatments
11. Has other primary cancer requiring treatment within the last 3 years, except for cervical intraepithelial neoplasia, ductal carcinoma in situ, or completely excised squamous or basal cell carcinoma
12. Is a pregnant or lactating female
13. Had major surgery, open biopsy, or significant traumatic injury within 4 weeks prior to the first dose of study treatment
14. Is receiving or has received any investigational treatment within 4 weeks prior to study entry, or participating in another clinical study
15. Has known DPD deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLT) and incidence of adverse events as assessed by CTCAE v5.0 | ~6 months
  Frequency, duration, and severity of DLTs and adverse events (AEs)
Maximum Plasma Concentration (Cmax) of capecitabine | ~14 days
  To evaluate the Maximum Plasma Concentration (Cmax) of capecitabine

SECONDARY OUTCOMES:
QTc effect of PCS6422 | ~6 months
  To evaluate the effect of PCS6422 on QTc
Maximum Plasma Concentration (Cmax) of PCS6422 | ~14 days
  To evaluate the Maximum Plasma Concentration (Cmax) of PCS6422
Number of participants with Adverse Events of Special Interest (AESI) | ~6 months
  Frequency, duration and severity of AESIs

CONTACTS AND LOCATIONS:
Overall Officials: Sian Bigora, Pharm. D, Study Director — Processa Pharmaceuticals
Locations (6):
- United States (6):
  - Processa Clinical Site, Omaha, Nebraska
  - Processa Clinical Site, New Brunswick, New Jersey
  - Processa Clinical Site, Santa Fe, New Mexico
  - Processa Clinical Site, New York, New York
  - Processa Clinical Site, Cleveland, Ohio
  - Processa Clinical Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No